CLINICAL TRIAL: NCT03999658
Title: An Open-label, Multicenter, Global Phase 2 Basket Study to Investigate the Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of STI-3031 in Patients With Selected Relapsed or Refractory Malignancies.
Brief Title: A Study of STI-3031 (an Anti-PD-L1 Antibody) in Patients With Selected Relapsed/Refractory Malignancies
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sorrento Therapeutics filed for chapter 11 bankruptcy.
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STI-3031-001
Record Dates: First submitted 2019-06-24; First posted 2019-06-27 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Peripheral T Cell Lymphoma; Diffuse Large B Cell Lymphoma; Biliary Tract Cancer; Extranodal NK T Cell Lymphoma, Nasal
Keywords: ENKTL; DLBCL; PTCL; cholangiocarcinoma; gall bladder cancer; relapsed; refractory; T/NK-cell; NK/T-cell; peripheral T-cell; PD-L1; anti-PD-L1 antibody
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, Large B-Cell, Diffuse; Biliary Tract Neoplasms; Lymphoma, Extranodal NK-T-Cell; Cholangiocarcinoma; Gallbladder Neoplasms; Recurrence | interventions — IMC-001

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Extranodal NK/T-cell lymphoma (ENKTL) (Experimental): Intravenous STI-3031 (anti-PD-L1 antibody)
  Interventions: Biological: STI-3031
- Peripheral T-cell lymphomas (PTCL) (Experimental): Intravenous STI-3031 (anti-PD-L1 antibody)
  Interventions: Biological: STI-3031
- Diffuse large B-cell lymphoma (DLBCL) (Experimental): Intravenous STI-3031 (anti-PD-L1 antibody)
  Interventions: Biological: STI-3031
- Biliary tract cancers (BTC) (Experimental): Intravenous STI-3031 (anti-PD-L1 antibody)
  Interventions: Biological: STI-3031

INTERVENTIONS:
Biological: STI-3031 — anti-PD-L1 antibody
  Other Names: IMC-001

SUMMARY:
This study evaluates the efficacy, as measured by the objective response rate, of STI-3031, an anti-PD-L1 antibody, in previously treated patients with selected advanced lymphomas or biliary tract cancer.

DETAILED DESCRIPTION:
This is an open-label, multicenter, global Phase 2 basket study to investigate the efficacy, safety, pharmacokinetics and pharmacodynamics of STI-3031 in patients with selected relapsed or refractory (R/R) malignancies. The study will be conducted as separate Phase 2, single arm substudies for each of the indications below:

* Extranodal NK/T-cell lymphoma (ENKTL)
* Peripheral T-cell lymphomas (PTCL)
* Diffuse large B-cell lymphoma (DLBCL) with PD-L1 gene translocation, copy gain, amplification, polysomy detectable by a fluorescence in situ hybridization (FISH) assay or Epstein-Barr virus positivity (EBV+) as assessed by EBV-encoded small RNA (EBER) testing
* Biliary tract cancers (BTC) (intrahepatic cholangiocarcinoma), extrahepatic cholangiocarcinoma or gallbladder cancer)

All participants will receive the study intervention, STI-3031.

ELIGIBILITY:
Inclusion Criteria:

* Documented histologically confirmed diagnoses of Extranodal NK/T-cell lymphoma, Peripheral T-cell lymphoma, Diffuse Large B-cell lymphoma (with a PD-L1 gene abnormality or Epstein-Barr virus positivity, or biliary tract cancer.
* Prior treatment:

  * Extranodal NK/T-cell lymphoma: Must have received at least 1 previous line of systemic therapy including an asparaginase-based regimen.
  * Peripheral T-cell lymphoma: must have received at least 1 previous line of systemic multi-agent chemotherapy. Participants with anaplastic large cell lymphoma (ALCL) must have received brentuximab vedotin
  * Diffuse Large B-cell lymphoma: Must have received at least 2 previous lines of systemic therapy including an anti-CD20 antibody
  * Biliary Tract Cancer: Must have received at least 1 previous line of systemic therapy including gemcitabine with or without platinum
* Documented disease progression during or after the last therapy
* If not previously treated with transplant, Investigator considers the participant ineligible for transplant
* Measurable disease
* Adult age (as defined by respective country) at time of signing informed consent form (ICF)
* Must be able to understand the nature of the study and provide a signed and dated, written ICF prior to any study-specific procedures, sample collections and analyses
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 or 1
* Prior radiotherapy is allowed if more than 14 days have elapsed since the end of treatment and radiopharmaceuticals are permitted if more than 8 weeks have elapsed since the end of treatment
* At least 14 days or 5 half-lives must have elapsed since the last chemotherapy, immunotherapy, biological or investigational therapy, and have recovered from toxicities associated with such treatment to < Grade 2
* Adequate hematologic, renal and hepatic function
* Females of childbearing potential (FCBP) must agree to use a reliable form of contraceptive during the study treatment period and for at least 90 days following the last dose of study intervention
* Male participants must agree to use barrier contraception (i.e., condoms) for the duration of the study and for at least 90 days after the last dose of study intervention
* Predicted life expectancy of at least 16 weeks

Exclusion Criteria:

* Current participation in another therapeutic clinical trial
* Prior treatment with an anti-PD-L1 or anti-PD-1 antibody
* Patients with symptomatic central nervous system (CNS) metastases unless considered adequately treated and controlled for at least 2 weeks
* Prior hematopoietic stem cell transplantation
* History of other previous cancer that would interfere with the determination of safety or efficacy
* Any active autoimmune disease or a documented history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications, except for participants with vitiligo, hormone replacement therapy for stable thyroid diseases and Type 1 diabetes mellitus
* Apparent active or latent tuberculosis (TB) infection
* Seropositive for or have active infection with hepatitis C virus (HCV), unless HCV viral load is below the limit of quantification and participant is on concurrent viral suppressive therapy
* Seropositive for or have active viral infection with hepatitis B virus (HBV), unless HBV viral load is below the limit of quantification and participant is on concurrent viral suppressive therapy
* Seropositive for or active viral infection with HIV, unless the following are met:

  * CD4+ T-cell (CD4+) counts ≥ 350 cells/uL; and
  * Participant has been on established antiretroviral therapy (ART) for at least 4 weeks prior to screening and have HIV viral load < 400 copies/mL; and
  * Participant has not had acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections within the past 12 months prior to screening
* Active infection (viral, bacterial, or fungal) requiring intravenous (IV) systemic therapy within 14 days
* Evidence of bleeding diathesis or coagulopathy.
* Significant proteinuria
* Conditions requiring chronic steroid use (> 10 mg/day of prednisone or equivalent).
* Recent history of attenuated viral vaccination within 30 days prior to the first dose of study intervention
* Herbal preparations/medications are not allowed throughout the treatment period unless first discussed with and approved by the Medical Monitor
* History of severe hypersensitivity reactions to other monoclonal antibodies or known hypersensitivity to the study intervention or its excipients.
* Known current drug or alcohol abuse
* Major surgical procedures ≤ 28 days prior to the first dose of study intervention, or minor surgical procedures ≤7 days prior to the first dose of study intervention
* Pregnant or lactating
* Any of the following cardiac diseases currently or within the last 6 months:

  * QT interval corrected using Fridericia's formula >450 milliseconds in men and > 470 milliseconds in women (up to 480 milliseconds may be allowed after discussion between the Investigator and the Medical Monitor).
  * Left Ventricular Ejection Fraction (LVEF) <45% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO)
  * Unstable angina pectoris
  * Congestive heart failure (New York Heart Association ≥ Grade 2)
  * Acute myocardial infarction
  * Clinically significant conduction abnormality not controlled with pacemaker or medication
  * Significant ventricular or supraventricular arrhythmias (Participants with chronic rate-controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible.)
* Underlying medical conditions that, in the opinion of the investigator and/or medical monitor, will render the administration of study drug hazardous or obscure the interpretation of safety or efficacy results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Approximately 24 months
  Percentage of participants achieving a Complete Response (CR) or Partial Response (PR) at any time during the study as assessed by an Independent Response Committee (IRC) per the Lugano criteria with LYRIC modification or RECIST 1.1

SECONDARY OUTCOMES:
Objective Response Rate by treating physician | Approximately 24 months
  Percentage of participants achieving a CR or PR at any time during the study as assessed by the Investigator per the Lugano criteria with LYRIC modification or RECIST 1.1
Duration of Response | Approximately 24 months
  Time from the first documentation of response (CR or PR) to the first documentation of progressive disease (PD) as assessed by an IRC per the Lugano criteria with LYRIC modification or RECIST 1.1
Complete Response Rate | Approximately 24 months
  Percentage of participants achieving a CR at any time during the study as assessed by an IRC per the Lugano criteria with LYRIC modification or RECIST 1.1
Duration of Complete Response Rate | Approximately 24 months
  Time from the first documentation of CR to the first documentation of PD as assessed by an IRC per the Lugano criteria with LYRIC modification or RECIST 1.1
Progressive-free survival | Approximately 24 months
  Time from enrollment until PD or death as assessed by an IRC per the Lugano criteria with LYRIC modification or RECIST 1.1
12-month Progressive-free survival | Approximately 30 months (18 months for enrollment plus 12 months follow-up for the last participant enrolled)
  Percentage of participants without PD or death at 12 months after their first dose of study intervention as assessed by an IRC per the Lugano criteria with LYRIC modification or RECIST 1.1
Event free survival | Approximately 24 months
  Time from enrollment to PD, death, or start of new treatment as assessed by an IRC per the Lugano criteria with LYRIC modification or RECIST 1.1
Area Under the Curve (AUC) of the blood levels of STI-3031 | Approximately 24 months
  Measure the actual body exposure to STI-3031
Maximum Plasma Concentration (Cmax) of STI-3031 | Approximately 24 months
  Measure the maximum (or peak) blood concentration of STI-3031
Time of Maximum concentration observed (Tmax) of STI-3031 | Approximately 24 months
  Measure the is the time at which the maximum blood concentration of STI-3031 is observed
Half-life (t1/2) of STI-3031 | Approximately 24 months
  Measure the time it takes for the concentration of the drug in the blood to be reduced by 50%
Immunogenicity | Approximately 24 months
  Incidence of anti-drug antibody (ADA) (serum titers of anti-STI-3031 antibodies) and correlation with exposure and activity
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of STI-3031 | Approximately 24 months
  Terms, frequency, severity and seriousness of adverse events (AEs) and relationship of AEs to STI-3031 the actual body exposure to drug after administration

IPD SHARING:
Plan to Share IPD: No